CLINICAL TRIAL: NCT03943953
Title: A Pilot Study Evaluating the Effectiveness of Information and Therapy Guides for Improving the Psychosocial Wellbeing of People With Facial Palsy.
Brief Title: Self-guided Psychosocial Intervention for Facial Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Matthew Hotton, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14110
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2022-08

CONDITIONS: Facial Palsy
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Intervention Model Description: One single group will be trialling a new self-guided psychological intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Facial Palsy - Trial of ITG (Experimental): In this arm of the trial individuals with facial palsy will trial the use of information and therapy guides over a 4-6 week period. They will complete measures at the start and end of this period.
  Interventions: Behavioral: Information and Therapy Guides

INTERVENTIONS:
Behavioral: Information and Therapy Guides — We have developed seven self-guided information and therapy guides (ITGs), for people with facial palsy and/or their friends or relatives. We have written these guides by drawing on interventions with a strong evidence-base in other populations, such as cognitive behavioural therapy, social skills training and acceptance and commitment therapy:
  1. Facial palsy: Coping with the early stages.
  2. Facial palsy: Coping with comments, questions and staring.
  3. Facial palsy: Communicating with confidence.
  4. Facial palsy: Managing anxiety.
  5. Facial palsy: Managing your mood.
  6. Facial palsy: Building your self-esteem.
  7. Facial palsy: Advice for friends, family and partners.

SUMMARY:
Facial palsy affects between 23 to 35 people per 100,000. As well as affecting an individual's appearance, it also can lead to difficulties with: eating, drinking, speaking, eyelid closure, pain and taste.

Facial palsy has been shown to have a significant impact on an individual's psychological wellbeing, including issues with anxiety, depression and low self-esteem. These elevated levels of distress have been thought to be partly due to the impact that facial palsy has on the face's ability to express emotions, which is a crucial aspect of face-to-face communication.

Although not researched yet in a facial palsy population, one type of psychological intervention that has been found to be effective at improving the psychosocial wellbeing of people with visible differences has been psychological self-help. With this in mind, the investigators have developed seven self-guided information and therapy guides (ITGs), for people with facial palsy and/or their friends or relatives. The investigators have written these guides by drawing on interventions with a strong evidence-base in other populations, such as cognitive behavioural therapy, social skills training and acceptance and commitment therapy:

1. Facial palsy: Coping with the early stages.
2. Facial palsy: Coping with comments, questions and staring.
3. Facial palsy: Communicating with confidence.
4. Facial palsy: Managing anxiety.
5. Facial palsy: Managing your mood.
6. Facial palsy: Building your self-esteem.
7. Facial palsy: Advice for friends, family and partners.

The investigators aim to evaluate the effectiveness, usability and acceptability of these guides to people with facial palsy and/or their friends, family and partners, by piloting their use over a 4-6 week period. Assessment of psychosocial wellbeing will be carried out before and after the 4-6 week period, while participants will be invited to provide usability and acceptability feedback on the guides after the 4-6 week period.

DETAILED DESCRIPTION:
Given that this study represents an initial pilot of the use of self-guided information and therapy guides for people with facial palsy (and/or their friends and relatives), all eligible participants will receive the intervention (i.e. there will be no control group). As a result, this study will have a repeated-measures design.

Eligible participants will be recruited by one of two means:

1. Face-to-face of recruitment of OUH NHS patients during clinics at the Oxford Facial Palsy Service
2. Recruitment of people with facial palsy, not under the care of the Oxford Facial Palsy Service, through relevant web and social media pages (e.g. the Facial Palsy UK Facebook page)

Potential participants who have expressed an interest in the study will be provided with an information sheet, and be invited to provide written consent. Participants recruited through the Oxford Facial Palsy Service will proved written consent via Survey Hero, either in clinic or remotely online at a later if they wish for longer time to consider their involvement in the study. Participants recruited through Facial Palsy UK/social media will provide written consent via Survey Hero.

Once participants have provided consent, they will be provided with an online screening questionnaire (in order to check for eligibility). Participants recruited in Oxford Facial Palsy Service clinics will complete the screening questionnaire on the researcher's laptop. Alternatively, if participants recruited in clinic wish to have more time to consider whether or not to participate, they will be able to complete online screening (and subsequent baseline assessments) remotely online. Participants recruited on social media will be emailed a link to the screening questionnaire.

Eligible participants will then be invited to complete baseline questionnaires:

People with facial palsy: Hospital Anxiety and Depression Scale; FACE-Q Satisfaction with appearance; FACE-Q Psychological function; FACE-Q Social function and Facial Disability Index. The Facial Disability Index will allow for control of improvement in facial palsy symptoms over time.

Friends, relatives and partners: Hospital Anxiety and Depression Scale and Adult Carer Quality of Life Questionnaire.

Like the screening questionnaires, written consent and baseline questionnaires will be completed online.

Eligible participants will then be administered the relevant self-guided information and therapy guide. For eligible carers/relatives this will be the guide entitled "Facial palsy: Advice for friends, family and partners". For eligible participants with facial palsy, this will be determined by their score on the screening questionnaire.

Participants will then utilise the guide over a period of four-to-six weeks. Half-way through the intervention period (after 2-3 weeks), they will receive an email reminding them to complete the guide and will be provided a web-link to complete a questionnaire, designed for the purpose of the current study, measuring the participants' ratings of acceptability and usability of the guides (participant satisfaction questionnaire).

At the end of the four-to-six week period, participants will be re-administered the baseline questionnaires, along with a questionnaire designed for the purpose of the current study measuring the participants' ratings of acceptability and usability of the guides (participant satisfaction questionnaire). Participants with facial palsy will also be re-administered the initial screening questionnaire. This will indicate whether the participant is eligible to complete a further guide. If this is the case, then their post-intervention questionnaires will serve as a new baseline and the participant will be invited to complete the new guide over a second four-to-six week period (followed by the same follow-up assessments as followed the first guide). This process will occur up to a maximum of six times (reflecting the potential for a participant to trial all six guides). If they do not wish to complete further guides then the participant will be thanked for their involvement in the study and their involvement will be registered as 'complete'.

Friends, relatives and partners of people with facial palsy will only be required to complete pre and post questionnaires if they are actively involved in the study due to completing the friend, relative or partner ITG. Likewise, individuals with facial palsy are not required to complete questionnaires if they are not actively involved in the study (i.e. not trialing and ITG), but their friend or relative is.

The investigators aim to trial the guides over a period of one year (May 2019 - May 2020). This will lead to the predicted sample size of 140 participants (120 with facial palsy, 20 per each of the 6 guides; 20 friends and family). This target is based on there being approximately 3000 people who have access to the Facial Palsy UK website. Given that approximately one-third of people with facial palsy experience a significant level of distress; the investigators hope that our guides would be relevant to, and accessible by, around 1000 people. 140 is therefore a conservative estimate of the number of participants that the investigators will be able to recruit.

Participants recruited from OUH NHS Foundation trust will be provided with an information sheet during their clinic appointment with the Oxford Facial Palsy Service. Written consent will be obtained in the clinic by a member of the research team.

Participants recruited from social media will be provided with an information sheet via email and will provide written consent online.

ELIGIBILITY:
Inclusion Criteria:

Participant with Facial Palsy:

* Participant is willing and able to give informed consent for participation in the study.
* Aged 18 years or above.
* Current diagnosis of facial palsy, of any severity or aetiology.
* Participants experience one or more psychosocial difficulties related to facial palsy 'all the time' or 'a lot of the time', as assessed by a screening questionnaire

Participant who is a friend, family member or partner of someone with facial palsy:

* Participant is willing and able to give informed consent for participation in the study.
* Aged 18 years or above.
* Is a friend, family member or partner of an adult with facial palsy, of any severity or aetiology.
* Participants experience psychosocial difficulties related to supporting someone with facial palsy, as assessed by participant responding 'all the time' or 'a lot of the time' to one or more questions on a screening questionnaire

Exclusion Criteria:

Participant with Facial Palsy:

* The participant is not in within the target age range (e.g. under the age of 18 years).
* They are not an individual with a current diagnosis of facial palsy.
* They do not speak enough English to understand the questionnaires or ITGs.
* They do not meet eligibility on the screening questionnaire (i.e. they 'never' or 'only occasionally' experience psychosocial difficulties associated with facial palsy (see section 7.2 Screening and Eligibility Assessment).

Participant who is a friend, family member or partner of someone with facial palsy:

* The participant is not in within the target age range (e.g. under the age of 18 years).
* They are not a friend, family member or partner of an adult with a current diagnosis of facial palsy.
* They do not speak enough English to understand the questionnaires or ITG.
* They do not meet eligibility on the screening questionnaire (i.e. they 'never' or 'only occasionally' experience psychosocial difficulties associated with supporting someone with facial palsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hotton, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, Oxon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to make data available

REFERENCES:
- [Background] Fu L, Bundy C, Sadiq SA. Psychological distress in people with disfigurement from facial palsy. Eye (Lond). 2011 Oct;25(10):1322-6. doi: 10.1038/eye.2011.158. Epub 2011 Jul 1. PMID 21720412
- [Background] Coulson SE, O'dwyer NJ, Adams RD, Croxson GR. Expression of emotion and quality of life after facial nerve paralysis. Otol Neurotol. 2004 Nov;25(6):1014-9. doi: 10.1097/00129492-200411000-00026. PMID 15547436
- [Background] Muftin Z, Thompson AR. A systematic review of self-help for disfigurement: effectiveness, usability, and acceptability. Body Image. 2013 Sep;10(4):442-50. doi: 10.1016/j.bodyim.2013.07.005. Epub 2013 Aug 17. PMID 23962642
- [Background] Martyn CN, Hughes RA. Epidemiology of peripheral neuropathy. J Neurol Neurosurg Psychiatry. 1997 Apr;62(4):310-8. doi: 10.1136/jnnp.62.4.310. No abstract available. PMID 9120441
- [Background] Hultcrantz M. Rehabilitation of Bells' palsy from a multi-team perspective. Acta Otolaryngol. 2016;136(4):363-7. doi: 10.3109/00016489.2015.1116124. Epub 2015 Dec 4. PMID 26634395
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Klassen AF, Cano SJ, Alderman A, East C, Badia L, Baker SB, Robson S, Pusic AL. Self-Report Scales to Measure Expectations and Appearance-Related Psychosocial Distress in Patients Seeking Cosmetic Treatments. Aesthet Surg J. 2016 Oct;36(9):1068-78. doi: 10.1093/asj/sjw078. Epub 2016 May 24. PMID 27222106
- [Background] VanSwearingen JM, Brach JS. The Facial Disability Index: reliability and validity of a disability assessment instrument for disorders of the facial neuromuscular system. Phys Ther. 1996 Dec;76(12):1288-98; discussion 1298-300. doi: 10.1093/ptj/76.12.1288. PMID 8959998
- [Derived] Hotton M, Johnson D, Kilcoyne S, Dalton L. Evaluating the effectiveness and acceptability of information and therapy guides for improving the psychosocial well-being of people with facial palsy. J Plast Reconstr Aesthet Surg. 2022 Sep;75(9):3356-3364. doi: 10.1016/j.bjps.2022.04.022. Epub 2022 Apr 25. PMID 35623976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The aim of this project was for participants to test a total of 140 Information and Therapy Guides. Because many participants were eligible to test multiple guides, the number of participants enrolled is lower than 140.
Groups:
- Facial Palsy - Trial of ITG: In this arm of the trial individuals with facial palsy will trial the use of information and therapy guides over a 4-6 week period. They will complete measures at the start and end of this period.
  Information and Therapy Guides: We have developed seven self-guided information and therapy guides (ITGs), for people with facial palsy and/or their friends or relatives. We have written these guides by drawing on interventions with a strong evidence-base in other populations, such as cognitive behavioural therapy, social skills training and acceptance and commitment therapy:
  1. Facial palsy: Coping with the early stages.
  2. Facial palsy: Coping with comments, questions and staring.
  3. Facial palsy: Communicating with confidence.
  4. Facial palsy: Managing anxiety.
  5. Facial palsy: Managing your mood.
  6. Facial palsy: Building your self-esteem.
- Friends and Family - ITG: In this arm of the trial friends and famileis of individuals with facial palsy will trial the use of information and therapy guides over a 4-6 week period. They will complete measures at the start and end of this period.
  Information and Therapy Guides: Facial palsy: Advice for friends, family and partners.
Period: Trial of ITG 1
Arm/Group | Facial Palsy - Trial of ITG | Friends and Family - ITG
Started | 88 (88 unique participants were enrolled at the outset. 44 of these were re-enrolled to trial a second guide. 18 of these re-enrolled to trial a third guide. 10 of these re-enrolled to trial a fourth guide. Three of these re-enrolled to trial a fifth guide. These 88 participants provided a total of 132 Time 1 data points) | 9
Completed | 69 (57 unique participants completed the study (e.g. completed all guides they had been enrolled to trial).) | 8
Not Completed | 19 | 1
Not completed — Lost to Follow-up | 19 | 1
Period: Trial of ITG 2
Arm/Group | Facial Palsy - Trial of ITG | Friends and Family - ITG
Started | 44 (The number of participants trialling a second guide was lower than the number trailling the first guide, as not all were eligible to trial a second guide) | 0 (There was only one ITG available to friends and family)
Completed | 36 | 0 (There was only one ITG available to friends and family)
Not Completed | 8 | 0
Not completed — Lost to Follow-up | 8 | 0
Period: Trial of ITG 3
Arm/Group | Facial Palsy - Trial of ITG | Friends and Family - ITG
Started | 18 (The number of participants trialling a third guide was lower than the number trailling the second guide, as not all were eligible to trial a further third guide) | 0
Completed | 16 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: Trial of ITG 4
Arm/Group | Facial Palsy - Trial of ITG | Friends and Family - ITG
Started | 10 (The number of participants trialling a fourth guide was lower than the number trailling the third guide, as not all were eligible to trial a further fourth guide) | 0
Completed | 8 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: Trial of ITG 5
Arm/Group | Facial Palsy - Trial of ITG | Friends and Family - ITG
Started | 3 (The number of participants trialling a fifth guide was lower than the number trailling the fourth guide, as not all were eligible to trial a further fifth guide) | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Facial Palsy - Trial of ITG: In this arm of the trial individuals with facial palsy will trial the use of information and therapy guides over a 4-6 week period. They will complete measures at the start and end of this period.
  Information and Therapy Guides: We have developed seven self-guided information and therapy guides (ITGs), for people with facial palsy and/or their friends or relatives. We have written these guides by drawing on interventions with a strong evidence-base in other populations, such as cognitive behavioural therapy, social skills training and acceptance and commitment therapy:
  1. Facial palsy: Coping with the early stages.
  2. Facial palsy: Coping with comments, questions and staring.
  3. Facial palsy: Communicating with confidence.
  4. Facial palsy: Managing anxiety.
  5. Facial palsy: Managing your mood.
  6. Facial palsy: Building your self-esteem.
  7. Facial palsy: Advice for friends, family and partners.
- Friends and Family - Trial of ITG: In this arm of the trial friends and family of individuals with facial palsy will trial the use of information and therapy guides over a 4-6 week period. They will complete measures at the start and end of this period.
  ITG: Facial palsy: Advice for friends, family and partners.
- Total: Total of all reporting groups
Arm/Group | Facial Palsy - Trial of ITG | Friends and Family - Trial of ITG | Total
Number analyzed (Participants) | 88 | 9 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.06 (13.62) | 45.00 (18.04) | 45.96 (14.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 2 | 85
  Male | 5 | 7 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 88 | 9 | 97
FACE-Q Psychological Function [Mean (Standard Deviation); unit: units on a scale] — This 10-item scale measures psychological wellbeing using a series of positively worded statements, with participants invited to rate how much they agree/disagree with each statement. There is a minimum score of 10 and a maximum score of 40. Scores are Rasch transformed to a 0-100 scale. A high score indicates greater psychological wellbeing. Population: Friends and family members did not complete this measure
  units on a scale
    number analyzed (Participants) | 88 | 0 | 88
    (all) | 38.19 (15.46) |  | 38.19 (15.46)
FACE-Q Social Function [Mean (Standard Deviation); unit: units on a scale] — In this scale there are 8 statements pertaining to measuring social functioning. Scores on this scale range from 8 to 32, with scores Rasch transformed to a 0-100 scale. Higher scores indicate better social function. Population: Friends and family members did not complete this measure at baseline
  units on a scale
    number analyzed (Participants) | 88 | 0 | 88
    (all) | 33.9 (18.37) |  | 33.9 (18.37)
Facial Disability Index (Social Function) [Mean (Standard Deviation); unit: units on a scale] — A 5-item self-report measure of social function in people with facial palsy. The scale is scored out of 100 (100 = high function). Population: Friends and family members did not complete this measure at baseline
  units on a scale
    number analyzed (Participants) | 88 | 0 | 88
    (all) | 49.15 (19.74) |  | 49.15 (19.74)
FACE-Q Appearance-Related Psychosocial Distress [Mean (Standard Deviation); unit: units on a scale] — An eight-item scale assessing an individual's concerns regarding their facial appearance on a scale of 8-32, which is then Rasch transformed to a 0-100 scale. The higher the score, the greater the patient's dissatisfaction with their appearance. Population: Friends and family members did not complete this measure at baseline
  units on a scale
    number analyzed (Participants) | 88 | 0 | 88
    (all) | 65.18 (15.53) |  | 65.18 (15.53)
Hospital Anxiety and Depression Scale [Mean (Standard Deviation); unit: units on a scale] — A 14-item scale with two seven-item subscales looking at anxiety and depression. A score equal-to-or-lower-than 7 on a subscale falls below the clinical cut-off, a score of 8-10 indicates probably clinically significant anxiety or depression, while a score of 11 or more indicates clinically significant anxiety or depression. Scores range from 0-52, with a higher score indicating higher severity. Population: Friends and family members did not complete this measure at baseline
  units on a scale | 18.01 (7.77) | 9.33 (5.05) | 17.20 (7.58)

OUTCOME MEASURES:

1. Primary Outcome: FACE-Q Psychological Function
Description: This 10-item scale measures psychological wellbeing using a series of positively worded statements, with participants invited to rate how much they agree/disagree with each statement. There is a minimum score of 10 and a maximum score of 40. Scores are Rasch transformed to a 0-100 scale. A high score indicates greater psychological wellbeing.
  As some participants were eligible to trial multiple guides, some participants contributed multiple data points.
Time Frame: Time 1: Baseline
Population: This measure was not collected for friends and family
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Data points
Arm/Group | Facial Palsy - Trial of ITG
Number analyzed (Participants) | 88
Number analyzed (Data points) | 132
units on a scale | 38.19 (15.46)

2. Primary Outcome: FACE-Q Psychological Function
Description: as for outcome 1
Time Frame: Time 2: 4-6 week follow-up
Population: This measure was not collected for friends and family
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Data points
Arm/Group | Facial Palsy - Trial of ITG
Number analyzed (Participants) | 88
Number analyzed (Data points) | 132
units on a scale | 41.05 (17.68)
Statistical Analysis 1: Comparison: Facial Palsy - Trial of ITG; This is a comparison between Time 1 and Time 2; Test type: Superiority; p = .018, t-test, 1 sided; Mean Difference (Final Values) = 2.86

3. Primary Outcome: FACE-Q Social Function
Description: In this scale there are 8 statements pertaining to measuring social functioning. Scores on this scale range from 8 to 32, with scores Rasch transformed to a 0-100 scale. Higher scores indicate better social function.
  As some participants were eligible to trial multiple guides, some participants contributed multiple data points.
Time Frame: Time 1: Baseline
Population: This measure was not collected for friends and family
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Data points
Arm/Group | Facial Palsy - Trial of ITG
Number analyzed (Participants) | 88
Number analyzed (Data points) | 132
units on a scale | 49.15 (18.34)

4. Primary Outcome: FACE-Q Social Function
Description: as for outcome 3
Time Frame: Time 2: 4-6 week follow-up
Population: This measure was not collected for friends and family
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Data points
Arm/Group | Facial Palsy - Trial of ITG
Number analyzed (Participants) | 88
Number analyzed (Data points) | 132
units on a scale | 53.03 (20.43)
Statistical Analysis 1: Comparison: Facial Palsy - Trial of ITG; This is a comparison between Time 1 and Time 2; Test type: Superiority; p = .001, t-test, 1 sided; Mean Difference (Final Values) = 3.88

5. Primary Outcome: Facial Disability Index (Social Function)
Description: A 5-item self-report measure of social function in people with facial palsy. The scale is scored out of 100 (100 = high function).
  As some participants were eligible to trial multiple guides, some participants contributed multiple data points.
Time Frame: Time 1: Baseline
Population: This measure was not collected for friends and family
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Data points
Arm/Group | Facial Palsy - Trial of ITG
Number analyzed (Participants) | 88
Number analyzed (Data points) | 132
units on a scale | 49.15 (19.74)

6. Primary Outcome: Facial Disability Index (Social Function)
Description: as for outcome 5
Time Frame: Time 2: 4-6 week follow-up
Population: This measure was not collected for friends and family
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Data points
Arm/Group | Facial Palsy - Trial of ITG
Number analyzed (Participants) | 88
Number analyzed (Data points) | 132
units on a scale | 53.03 (20.43)
Statistical Analysis 1: Comparison: Facial Palsy - Trial of ITG; This is a comparison between Time 1 and Time 2; Test type: Superiority; p = .006, t-test, 1 sided; Mean Difference (Final Values) = 3.88

7. Primary Outcome: FACE-Q Appearance-Related Psychosocial Distress
Description: An eight-item scale assessing an individual's concerns regarding their facial appearance on a scale of 8-32, which is then Rasch transformed to a 0-100 scale. The higher the score, the greater the patient's dissatisfaction with their appearance.
  As some participants were eligible to trial multiple guides, some participants contributed multiple data points.
Time Frame: Time 1: Baseline
Population: This measure was not collected for friends and family
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Data points
Arm/Group | Facial Palsy - Trial of ITG
Number analyzed (Participants) | 88
Number analyzed (Data points) | 132
units on a scale | 65.18 (15.53)

8. Primary Outcome: FACE-Q Appearance-Related Psychosocial Distress
Description: as for outcome 7
Time Frame: Time 2: 4-6 week follow-up
Population: This measure was not collected for friends and family
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Data points
Arm/Group | Facial Palsy - Trial of ITG
Number analyzed (Participants) | 88
Number analyzed (Data points) | 132
units on a scale | 62.90 (15.03)
Statistical Analysis 1: Comparison: Facial Palsy - Trial of ITG; This is a comparison between Time 1 and Time 2; Test type: Superiority; p = .035, t-test, 1 sided; Mean Difference (Final Values) = -2.28

9. Primary Outcome: Hospital Anxiety and Depression Scale
Description: A 14-item scale with two seven-item subscales looking at anxiety and depression. A score equal-to-or-lower-than 7 on a subscale falls below the clinical cut-off, a score of 8-10 indicates probably clinically significant anxiety or depression, while a score of 11 or more indicates clinically significant anxiety or depression. Scores range from 0-52, with a higher score indicating higher severity.
  As some participants with facial palsy were eligible to trial multiple guides, some participants with facial palsy contributed multiple data points.
Time Frame: Time 1: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Data points
Groups:
- Friends and Family: Friends, family members and carers
Arm/Group | Facial Palsy - Trial of ITG | Friends and Family
Number analyzed (Participants) | 88 | 8
Number analyzed (Data points) | 132 | 8
units on a scale | 18.01 (7.77) | 10.00 (4.96)

10. Primary Outcome: Hospital Anxiety and Depression Scale
Description: as for outcome 9
Time Frame: Time 2: 4-6 week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Data points
Groups:
- Friends and Family: Friends, family and carers of people with facial palsy
Arm/Group | Facial Palsy - Trial of ITG | Friends and Family
Number analyzed (Participants) | 88 | 8
Number analyzed (Data points) | 132 | 8
units on a scale | 17.61 (8.12) | 9.25 (4.65)
Statistical Analysis 1: Comparison: Facial Palsy - Trial of ITG; This is a comparison between Time 1 and Time 2; Test type: Superiority; p = .39, t-test, 1 sided; Mean Difference (Final Values) = -0.40

11. Secondary Outcome: Adult Carer Quality of Life Questionnaire
Description: 40 item questionnaire assessing carer quality of life. Possible scores range from 0-120, with higher scores indicating higher quality of life
Time Frame: Time 1: Baseline
Population: This measure was not collected for people with facial palsy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Friends and Family - ITG
Number analyzed (Participants) | 8
units on a scale | 56.88 (10.02)

12. Secondary Outcome: Adult Carer Quality of Life Questionnaire
Description: as for outcome 11
Time Frame: Time 2: 4-6 week follow-up
Population: This measure was not collected for people with facial palsy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Friends and Family - ITG
Number analyzed (Participants) | 8
units on a scale | 64.88 (10.06)

ADVERSE EVENTS:
Time Frame: Four to six weeks
Groups:
- Friends and Family: Friends, family and carers of people with facial palsy, testing the guide: Facial palsy: Advice for friends, family and partners.
Arm/Group | Facial Palsy - Trial of ITG | Friends and Family
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/9
Other Adverse Events (participants affected / at risk) | 0/88 | 0/9

LIMITATIONS AND CAVEATS:
* Over representation of female participants
* Small number of participants trialling each guide meant guides were evaluated collectively
* 31 participants were lost to follow-up, partly due to the suspension of the trial due to Covid-19
* No randomisation or control group was included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT03943953/Prot_SAP_000.pdf